CLINICAL TRIAL: NCT04232137
Title: Traditional Ethiopian Coffee Ceremony in a Rural Ethiopian Hospital to Increase Hospital-based Delivery Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Gambo General Rural Hospital (Other); University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Tobias Limperg, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GH/LUC/909
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Birth Setting; Maternal Health
Keywords: Coffee ceremony; Hospital-based deliveries; Maternal health; Ethiopia

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coffee ceremony (Experimental): Antenatal care patients will be told on their first antenatal care visit that a postpartum coffee ceremony will be organized for them and up to 4 relatives
  Interventions: Behavioral: Postpartum coffee ceremony
- NO Coffee ceremony (No Intervention): Antenatal care patients will be told that they will NOT receive a postpartum coffee ceremony, as is the current status quo

INTERVENTIONS:
Behavioral: Postpartum coffee ceremony — The promise of a postpartum coffee ceremony
  Arms: Coffee ceremony

SUMMARY:
This study evaluates if organizing a postpartum traditional Ethiopian coffee ceremony will provide an incentive for our antenatal care patients to eventually deliver in our hospital. Patients are randomized to either receiving, or not receiving, a postpartum coffee ceremony for them and their relatives.

DETAILED DESCRIPTION:
Ethiopia has one of the highest maternal mortality rates in the world, with an estimated maternal mortality ratio of 497 per 100,000 live births. Cultural factors contribute to the underutilization of maternal health services. In 2014, only 20% of our antenatal care patients delivered in our hospital. In order to increase health facility-based delivery rates, government-funded hospitals and health centers facilitate traditional Ethiopian coffee ceremonies after delivery. We hypothesized that organizing postpartum coffee ceremonies would motivate our antenatal care patients to deliver in our hospital and would thus increase the hospital-based delivery rate.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patient
* First visit to antenatal care clinic

Exclusion Criteria:

* Non-viable pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Limperg, MD MSc, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: Yes
All collected individual deidentified participant data will be shared.
Supporting Information: Study Protocol
Time Frame: Plan: immediately following publication. End date to be determined.
Access Criteria: Anyone who wishes to access the data. For any type of purpose.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Coffee Ceremony | NO Coffee Ceremony
Started | 254 | 185
Completed | 254 | 185
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coffee Ceremony | NO Coffee Ceremony | Total
Number analyzed (Participants) | 237 | 167 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (5.3) | 25.5 (5.5) | 25 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237 | 167 | 404
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Oromo | 226 | 155 | 381
  Other | 27 | 26 | 53
  Missing | 1 | 4 | 5
Antenatal care visits [Mean (Standard Deviation); unit: visits] | 1.75 (1) | 1.73 (1) | 1.74 (1)
Travel time to hospital [Mean (Standard Deviation); unit: minutes] | 100.7 (53) | 103.5 (52.2) | 101.9 (52.6)
Cost of transportation [Mean (Standard Deviation); unit: Ethiopian birr] | 6.2 (10.3) | 6.9 (13.3) | 6.5 (11.6)
Religion [Count of Participants; unit: Participants]
  Muslim | 198 | 137 | 335
  Other | 37 | 27 | 64
  Missing | 2 | 3 | 5
Education grade [Mean (Standard Deviation); unit: grades] | 5 (3.9) | 5.3 (3.9) | 5.1 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Hospital-based Delivery Rate
Description: Percentage of antenatal care patients that deliver in the hospital
Time Frame: Up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Coffee Ceremony | NO Coffee Ceremony
Number analyzed (Participants) | 237 | 167
Participants | 76 | 53

2. Secondary Outcome: Health Center or Health Post-delivery Rate
Description: Percentage of antenatal care patients that deliver in an associated health center or health post
Time Frame: Up to 9 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Coffee Ceremony | NO Coffee Ceremony
Serious Adverse Events (participants affected / at risk) | 0/237 | 0/167
Other Adverse Events (participants affected / at risk) | 0/237 | 0/167

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No